CLINICAL TRIAL: NCT02970123
Title: Sit Less, Interact, Move More (SLIMM) Intervention for Sedentary Behavior in Chronic Kidney Disease (CKD)
Acronym: SLIMM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Srinvasan Beddhu (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Srinvasan Beddhu, Principal Investigator, University of Utah
Organization: University of Utah (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB_00093477; 1R21DK106574-01A1 (NIH)
Record Dates: First submitted 2016-11-17; First posted 2016-11-21 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SLIMM Intervention (Experimental): Sit Less, Interact, Move More (SLIMM): instruction and monitoring feedback to promote decrease in sedentary activity duration, increase in casual walking duration, and increase in sedentary breaks
  Interventions: Behavioral: Sit Less, Interact, Move More (SLIMM)
- Standard of Care (No Intervention): Subjects will receive standard of care treatment for chronic kidney disease, with no instruction or feedback to alter sedentary or casual walking durations

INTERVENTIONS:
Behavioral: Sit Less, Interact, Move More (SLIMM)
  Arms: SLIMM Intervention

SUMMARY:
Sedentary behavior is engaging in activities in the seated or lying position that barely raise the energy expenditure level and has emerged as an important risk factor for obesity, diabetes, cardiovascular disease and mortality.

The primary hypothesis is that the Sit Less, Interact, Move More (SLIMM) intervention in Chronic Kidney Disease (CKD) will be effective in decreasing sedentary duration by increasing casual walking duration and thereby, increase physical activity energy expenditure.

DETAILED DESCRIPTION:
There are an estimated 15.5 million adults with stage 3 chronic kidney disease (CKD) while only about 600,000 patients have end-stage renal disease (ESRD) in the United States. This is because most of the people with CKD die before they reach ESRD. In order to decrease the high mortality in the CKD population, the "non-renal" issues that contribute to increased morbidity and mortality in this population need to be addressed.

Relevance of sedentary behavior in CKD: Prolonged sitting time (as assessed by a questionnaire or television viewing time) was associated with lower kidney function. Total and light physical activities, measured objectively with an accelerometer were found to be positively associated with kidney function in a study of community dwelling adults. In an analysis of National Health and Nutrition Examination Survey (NHANES) data, it was noted that participants with CKD spent more than two-thirds of the awake time in sedentary activities and longer sedentary duration was associated with increased mortality. It was also noted in another study that compared to those with CKD, those on maintenance hemodialysis had 3.4 fold higher odds of being sedentary independent of demographics, co-morbidity, body size, serum C-Reactive Protein (CRP) and albumin. Thus, sedentary behavior is very common in CKD, appears to worsen with more advanced kidney failure and increases mortality risk in this population.

Feasibility of replacing sedentary activities with moderate/ vigorous physical activities: Moderate/ vigorous physical activities are less likely to be an effective replacement for sedentary activities as most Americans do not reach even the current goals and achieving the currently recommended levels of 2.5 hrs/ week of moderate/ vigorous activities would account only for 2% of the total awake time (112 hours/week). Therefore, decreasing sedentary activities must involve an increase in activities that are less intensive than moderate/ vigorous activities.

The concept of Non- Exercise Activity Thermogenesis (NEAT) and biological relevance of light intensity activity: In a overfeeding study, it was demonstrated that increase (average 336 kcal/day) in non- exercise activity thermogenesis accounted for 10-fold differences in fat storage, directly predicted resistance to fat gain and explained most of the variations in weight gain between participants. Obese persons have less non-exercise activity thermogenesis and spend an average of 2 hrs/d more in a seated position compared to lean persons. Objectively measured light activity was inversely associated with insulin resistance and cardiometabolic risk factors. Daily lifestyle activities were negatively associated with insulin resistance. Thus, replacing sedentary activities with non-exercise intensity activities of daily living could increase energy expenditure and decrease adiposity.

Determining what kind of light activity would be most beneficial in replacing sedentary activity: As standing (~ 1.5 Metabolic Equivalents of Task (METs)) is by definition non-sedentary (i.e. not sitting or lying down), one might consider replacing sitting duration with standing duration in order to decrease sedentary behavior. However, replacing sitting duration with casual walking (2 to 2.9 METs) duration might be even more beneficial. This notion is supported by the following theoretical calculations of energy expenditure. Assuming 16 hrs/day of awake time, it was calculated that the weekly energy expenditure for a person weighing 80 kg for trade-off of 1 to 5 min/hr of sedentary activity at 1.2 METs with 1.5 METs (standing intensity activities) or 2.5 METs (casual walking intensity activities). Additional kcal/week was calculated as the difference in energy expenditure between sedentary activity and 1.5 or 2.5 METs activity using the equation Kcal/ week = (METs/hr) x weight in kg X weekly duration of the physical activity. Trade-off of 1-5 min/hr of sedentary duration with standing intensity activities duration is expected to result in additional weekly expenditure of 50-250 Kcal only. On the other hand, similar trade off of sedentary duration with casual walking intensity activities duration is expected to result in ~ 200 to 1000 Kcal/ week of additional energy expenditure. This is consistent with prior observation that increase in non-exercise activities could lead to an additional 350 Kcal/d of energy expenditure in obese individuals.

Indeed, in the NHANES analyses, it was noted that trade-off sedentary duration for light intensity (2.0 to 2.9 METs) activities but not for very light intensity (1.5 to 1.9 METs) duration was associated with significantly lower risk of mortality. Thus, replacing sedentary duration with casual walking duration could increase energy expenditure and decrease mortality in CKD.

ELIGIBILITY:
Inclusion Criteria:

* Stage 3/4 Chronic Kidney Disease, as defined by estimated glomerular filtration rate (eGFR) 15 to < 60 ml/min/1.73m^2
* Body Mass Index (BMI): 25 to 39.9 kg/m^2
* Able to achieve gait speed of > 1 m/sec and able to walk ≥ 320 meters in the 6-minute walk test

Exclusion Criteria:

* Previous renal replacement therapy
* Life expectancy < 1 year
* Pregnancy
* Prison incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-09-12 (Actual); Study Completion 2019-09-12 (Actual)

PRIMARY OUTCOMES:
Change in Sedentary Activity Duration | Baseline and 24 Weeks
  Change in sedentary activity duration (average sedentary minutes per hour), as measured by a validated accelerometry monitor from baseline to 24 weeks
Change in Casual Walking Duration | Baseline and 24 Weeks
  Change in casual walking activity duration (average walking minutes per hour), as measured by a validated accelerometry monitor from baseline to 24 weeks

SECONDARY OUTCOMES:
Change in Waist Circumference | Baseline and 24 Weeks
  Change in waist circumference, measured in centimeters, from baseline to 24 weeks
Change in Non-Exercise Activity Thermogenesis | Baseline and 24 Weeks
  Change in non-exercise activity thermogenesis, measured in kilocalorie/kilogram/hour, from baseline to 24 weeks
Change in Physical Function | Baseline and 24 Weeks
  Change in walking distance, measured in meters, using the 6-minute walk test from baseline to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Srinivasan Beddhu, M.D., Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alhassan S, Lyden K, Howe C, Kozey Keadle S, Nwaokelemeh O, Freedson PS. Accuracy of accelerometer regression models in predicting energy expenditure and METs in children and youth. Pediatr Exerc Sci. 2012 Nov;24(4):519-36. doi: 10.1123/pes.24.4.519. PMID 23196761
- [Background] Freedson PS, Lyden K, Kozey-Keadle S, Staudenmayer J. Evaluation of artificial neural network algorithms for predicting METs and activity type from accelerometer data: validation on an independent sample. J Appl Physiol (1985). 2011 Dec;111(6):1804-12. doi: 10.1152/japplphysiol.00309.2011. Epub 2011 Sep 1. PMID 21885802
- [Background] Kozey SL, Lyden K, Howe CA, Staudenmayer JW, Freedson PS. Accelerometer output and MET values of common physical activities. Med Sci Sports Exerc. 2010 Sep;42(9):1776-84. doi: 10.1249/MSS.0b013e3181d479f2. PMID 20142781
- [Background] Kozey-Keadle S, Staudenmayer J, Libertine A, Mavilia M, Lyden K, Braun B, Freedson P. Changes in sedentary time and physical activity in response to an exercise training and/or lifestyle intervention. J Phys Act Health. 2014 Sep;11(7):1324-33. doi: 10.1123/jpah.2012-0340. Epub 2013 Oct 31. PMID 24184493
- [Background] Lyden K, Keadle SK, Staudenmayer J, Freedson PS. A method to estimate free-living active and sedentary behavior from an accelerometer. Med Sci Sports Exerc. 2014 Feb;46(2):386-97. doi: 10.1249/MSS.0b013e3182a42a2d. PMID 23860415
- [Background] Lyden K, Kozey Keadle SL, Staudenmayer JW, Freedson PS. Validity of two wearable monitors to estimate breaks from sedentary time. Med Sci Sports Exerc. 2012 Nov;44(11):2243-52. doi: 10.1249/MSS.0b013e318260c477. PMID 22648343
- [Background] Lyden K, Kozey SL, Staudenmeyer JW, Freedson PS. A comprehensive evaluation of commonly used accelerometer energy expenditure and MET prediction equations. Eur J Appl Physiol. 2011 Feb;111(2):187-201. doi: 10.1007/s00421-010-1639-8. Epub 2010 Sep 15. PMID 20842375
- [Background] Beddhu S, Wei G, Marcus RL, Chonchol M, Greene T. Light-intensity physical activities and mortality in the United States general population and CKD subpopulation. Clin J Am Soc Nephrol. 2015 Jul 7;10(7):1145-53. doi: 10.2215/CJN.08410814. Epub 2015 Apr 30. PMID 25931456
- [Background] Ryan CG, Grant PM, Tigbe WW, Granat MH. The validity and reliability of a novel activity monitor as a measure of walking. Br J Sports Med. 2006 Sep;40(9):779-84. doi: 10.1136/bjsm.2006.027276. Epub 2006 Jul 6. PMID 16825270
- [Background] Dowd KP, Harrington DM, Donnelly AE. Criterion and concurrent validity of the activPAL professional physical activity monitor in adolescent females. PLoS One. 2012;7(10):e47633. doi: 10.1371/journal.pone.0047633. Epub 2012 Oct 19. PMID 23094069
- [Background] Harrington DM, Welk GJ, Donnelly AE. Validation of MET estimates and step measurement using the ActivPAL physical activity logger. J Sports Sci. 2011 Mar;29(6):627-33. doi: 10.1080/02640414.2010.549499. PMID 21360402
- [Background] Ainsworth BE, Haskell WL, Herrmann SD, Meckes N, Bassett DR Jr, Tudor-Locke C, Greer JL, Vezina J, Whitt-Glover MC, Leon AS. 2011 Compendium of Physical Activities: a second update of codes and MET values. Med Sci Sports Exerc. 2011 Aug;43(8):1575-81. doi: 10.1249/MSS.0b013e31821ece12. PMID 21681120
- [Background] Hu FB. Sedentary lifestyle and risk of obesity and type 2 diabetes. Lipids. 2003 Feb;38(2):103-8. doi: 10.1007/s11745-003-1038-4. PMID 12733740
- [Background] Freak-Poli R, Wolfe R, Peeters A. Risk of cardiovascular disease and diabetes in a working population with sedentary occupations. J Occup Environ Med. 2010 Nov;52(11):1132-7. doi: 10.1097/JOM.0b013e3181f8da77. PMID 21063192
- [Background] Hu FB, Li TY, Colditz GA, Willett WC, Manson JE. Television watching and other sedentary behaviors in relation to risk of obesity and type 2 diabetes mellitus in women. JAMA. 2003 Apr 9;289(14):1785-91. doi: 10.1001/jama.289.14.1785. PMID 12684356
- [Background] Pinto Pereira SM, Ki M, Power C. Sedentary behaviour and biomarkers for cardiovascular disease and diabetes in mid-life: the role of television-viewing and sitting at work. PLoS One. 2012;7(2):e31132. doi: 10.1371/journal.pone.0031132. Epub 2012 Feb 9. PMID 22347441
- [Background] Solomon TP, Thyfault JP. Type 2 diabetes sits in a chair. Diabetes Obes Metab. 2013 Nov;15(11):987-92. doi: 10.1111/dom.12105. Epub 2013 Apr 22. PMID 23551885
- [Background] Dunstan DW, Thorp AA, Healy GN. Prolonged sitting: is it a distinct coronary heart disease risk factor? Curr Opin Cardiol. 2011 Sep;26(5):412-9. doi: 10.1097/HCO.0b013e3283496605. PMID 21785350
- [Background] Hamilton MT, Hamilton DG, Zderic TW. Role of low energy expenditure and sitting in obesity, metabolic syndrome, type 2 diabetes, and cardiovascular disease. Diabetes. 2007 Nov;56(11):2655-67. doi: 10.2337/db07-0882. Epub 2007 Sep 7. PMID 17827399
- [Background] Henson J, Yates T, Edwardson CL, Khunti K, Talbot D, Gray LJ, Leigh TM, Carter P, Davies MJ. Sedentary time and markers of chronic low-grade inflammation in a high risk population. PLoS One. 2013 Oct 29;8(10):e78350. doi: 10.1371/journal.pone.0078350. eCollection 2013. PMID 24205208
- [Background] Thorp AA, Owen N, Neuhaus M, Dunstan DW. Sedentary behaviors and subsequent health outcomes in adults a systematic review of longitudinal studies, 1996-2011. Am J Prev Med. 2011 Aug;41(2):207-15. doi: 10.1016/j.amepre.2011.05.004. PMID 21767729
- [Background] Young DR, Reynolds K, Sidell M, Brar S, Ghai NR, Sternfeld B, Jacobsen SJ, Slezak JM, Caan B, Quinn VP. Effects of physical activity and sedentary time on the risk of heart failure. Circ Heart Fail. 2014 Jan;7(1):21-7. doi: 10.1161/CIRCHEARTFAILURE.113.000529. PMID 24449810
- [Background] Owen N, Healy GN, Matthews CE, Dunstan DW. Too much sitting: the population health science of sedentary behavior. Exerc Sport Sci Rev. 2010 Jul;38(3):105-13. doi: 10.1097/JES.0b013e3181e373a2. PMID 20577058
- [Background] Koster A, Caserotti P, Patel KV, Matthews CE, Berrigan D, Van Domelen DR, Brychta RJ, Chen KY, Harris TB. Association of sedentary time with mortality independent of moderate to vigorous physical activity. PLoS One. 2012;7(6):e37696. doi: 10.1371/journal.pone.0037696. Epub 2012 Jun 13. PMID 22719846
- [Background] Dunstan DW, Barr EL, Healy GN, Salmon J, Shaw JE, Balkau B, Magliano DJ, Cameron AJ, Zimmet PZ, Owen N. Television viewing time and mortality: the Australian Diabetes, Obesity and Lifestyle Study (AusDiab). Circulation. 2010 Jan 26;121(3):384-91. doi: 10.1161/CIRCULATIONAHA.109.894824. Epub 2010 Jan 11. PMID 20065160
- [Background] Tucker JM, Welk GJ, Beyler NK. Physical activity in U.S.: adults compliance with the Physical Activity Guidelines for Americans. Am J Prev Med. 2011 Apr;40(4):454-61. doi: 10.1016/j.amepre.2010.12.016. PMID 21406280
- [Background] Akber A, Portale AA, Johansen KL. Pedometer-assessed physical activity in children and young adults with CKD. Clin J Am Soc Nephrol. 2012 May;7(5):720-6. doi: 10.2215/CJN.06330611. Epub 2012 Mar 15. PMID 22422539
- [Background] Bharakhada N, Yates T, Davies MJ, Wilmot EG, Edwardson C, Henson J, Webb D, Khunti K. Association of sitting time and physical activity with CKD: a cross-sectional study in family practices. Am J Kidney Dis. 2012 Oct;60(4):583-90. doi: 10.1053/j.ajkd.2012.04.024. Epub 2012 Jun 19. PMID 22717340
- [Background] Hawkins MS, Sevick MA, Richardson CR, Fried LF, Arena VC, Kriska AM. Association between physical activity and kidney function: National Health and Nutrition Examination Survey. Med Sci Sports Exerc. 2011 Aug;43(8):1457-64. doi: 10.1249/MSS.0b013e31820c0130. PMID 21200336
- [Background] Coresh J, Selvin E, Stevens LA, Manzi J, Kusek JW, Eggers P, Van Lente F, Levey AS. Prevalence of chronic kidney disease in the United States. JAMA. 2007 Nov 7;298(17):2038-47. doi: 10.1001/jama.298.17.2038. PMID 17986697
- [Background] Anderton N, Giri A, Wei G, Marcus RL, Chen X, Bjordahl T, Habib A, Herrera J, Beddhu S. Sedentary Behavior in Individuals With Diabetic Chronic Kidney Disease and Maintenance Hemodialysis. J Ren Nutr. 2015 Jul;25(4):364-70. doi: 10.1053/j.jrn.2015.01.018. Epub 2015 Mar 5. PMID 25753603
- [Background] Troiano RP, Berrigan D, Dodd KW, Masse LC, Tilert T, McDowell M. Physical activity in the United States measured by accelerometer. Med Sci Sports Exerc. 2008 Jan;40(1):181-8. doi: 10.1249/mss.0b013e31815a51b3. PMID 18091006
- [Background] Levine JA, Eberhardt NL, Jensen MD. Role of nonexercise activity thermogenesis in resistance to fat gain in humans. Science. 1999 Jan 8;283(5399):212-4. doi: 10.1126/science.283.5399.212. PMID 9880251
- [Background] Levine JA, Lanningham-Foster LM, McCrady SK, Krizan AC, Olson LR, Kane PH, Jensen MD, Clark MM. Interindividual variation in posture allocation: possible role in human obesity. Science. 2005 Jan 28;307(5709):584-6. doi: 10.1126/science.1106561. PMID 15681386
- [Background] Healy GN, Dunstan DW, Salmon J, Cerin E, Shaw JE, Zimmet PZ, Owen N. Objectively measured light-intensity physical activity is independently associated with 2-h plasma glucose. Diabetes Care. 2007 Jun;30(6):1384-9. doi: 10.2337/dc07-0114. Epub 2007 May 1. PMID 17473059
- [Background] Healy GN, Wijndaele K, Dunstan DW, Shaw JE, Salmon J, Zimmet PZ, Owen N. Objectively measured sedentary time, physical activity, and metabolic risk: the Australian Diabetes, Obesity and Lifestyle Study (AusDiab). Diabetes Care. 2008 Feb;31(2):369-71. doi: 10.2337/dc07-1795. Epub 2007 Nov 13. PMID 18000181
- [Background] Nelson RK, Horowitz JF, Holleman RG, Swartz AM, Strath SJ, Kriska AM, Richardson CR. Daily physical activity predicts degree of insulin resistance: a cross-sectional observational study using the 2003-2004 National Health and Nutrition Examination Survey. Int J Behav Nutr Phys Act. 2013 Jan 28;10:10. doi: 10.1186/1479-5868-10-10. PMID 23351329
- [Background] Otten JJ, Jones KE, Littenberg B, Harvey-Berino J. Effects of television viewing reduction on energy intake and expenditure in overweight and obese adults: a randomized controlled trial. Arch Intern Med. 2009 Dec 14;169(22):2109-15. doi: 10.1001/archinternmed.2009.430. PMID 20008695
- [Background] Gardiner PA, Eakin EG, Healy GN, Owen N. Feasibility of reducing older adults' sedentary time. Am J Prev Med. 2011 Aug;41(2):174-7. doi: 10.1016/j.amepre.2011.03.020. PMID 21767725
- [Background] De Greef KP, Deforche BI, Ruige JB, Bouckaert JJ, Tudor-Locke CE, Kaufman JM, De Bourdeaudhuij IM. The effects of a pedometer-based behavioral modification program with telephone support on physical activity and sedentary behavior in type 2 diabetes patients. Patient Educ Couns. 2011 Aug;84(2):275-9. doi: 10.1016/j.pec.2010.07.010. Epub 2010 Aug 21. PMID 20732776
- [Background] Wellen KE, Hotamisligil GS. Inflammation, stress, and diabetes. J Clin Invest. 2005 May;115(5):1111-9. doi: 10.1172/JCI25102. PMID 15864338
- [Background] Greenberg AS, Obin MS. Obesity and the role of adipose tissue in inflammation and metabolism. Am J Clin Nutr. 2006 Feb;83(2):461S-465S. doi: 10.1093/ajcn/83.2.461S. PMID 16470013
- [Background] Anand S, Chertow GM, Johansen KL, Grimes B, Kurella Tamura M, Dalrymple LS, Kaysen GA. Association of self-reported physical activity with laboratory markers of nutrition and inflammation: the Comprehensive Dialysis Study. J Ren Nutr. 2011 Nov;21(6):429-37. doi: 10.1053/j.jrn.2010.09.007. Epub 2011 Jan 15. PMID 21239185
- [Background] Matsuzawa R, Matsunaga A, Wang G, Kutsuna T, Ishii A, Abe Y, Takagi Y, Yoshida A, Takahira N. Habitual physical activity measured by accelerometer and survival in maintenance hemodialysis patients. Clin J Am Soc Nephrol. 2012 Dec;7(12):2010-6. doi: 10.2215/CJN.03660412. Epub 2012 Sep 13. PMID 22977216
- [Background] Beddhu S, Baird BC, Zitterkoph J, Neilson J, Greene T. Physical activity and mortality in chronic kidney disease (NHANES III). Clin J Am Soc Nephrol. 2009 Dec;4(12):1901-6. doi: 10.2215/CJN.01970309. Epub 2009 Oct 9. PMID 19820134
- [Background] Fried LF, Lee JS, Shlipak M, Chertow GM, Green C, Ding J, Harris T, Newman AB. Chronic kidney disease and functional limitation in older people: health, aging and body composition study. J Am Geriatr Soc. 2006 May;54(5):750-6. doi: 10.1111/j.1532-5415.2006.00727.x. PMID 16696739
- [Background] Roshanravan B, Robinson-Cohen C, Patel KV, Ayers E, Littman AJ, de Boer IH, Ikizler TA, Himmelfarb J, Katzel LI, Kestenbaum B, Seliger S. Association between physical performance and all-cause mortality in CKD. J Am Soc Nephrol. 2013 Apr;24(5):822-30. doi: 10.1681/ASN.2012070702. Epub 2013 Apr 18. PMID 23599380
- [Background] Johansen KL, Kaysen GA, Dalrymple LS, Grimes BA, Glidden DV, Anand S, Chertow GM. Association of physical activity with survival among ambulatory patients on dialysis: the Comprehensive Dialysis Study. Clin J Am Soc Nephrol. 2013 Feb;8(2):248-53. doi: 10.2215/CJN.08560812. Epub 2012 Nov 2. PMID 23124787
- [Background] Sietsema KE, Amato A, Adler SG, Brass EP. Exercise capacity as a predictor of survival among ambulatory patients with end-stage renal disease. Kidney Int. 2004 Feb;65(2):719-24. doi: 10.1111/j.1523-1755.2004.00411.x. PMID 14717947
- [Background] Headley S, Germain M, Milch C, Pescatello L, Coughlin MA, Nindl BC, Cornelius A, Sullivan S, Gregory S, Wood R. Exercise training improves HR responses and V O2peak in predialysis kidney patients. Med Sci Sports Exerc. 2012 Dec;44(12):2392-9. doi: 10.1249/MSS.0b013e318268c70c. PMID 22811032
- [Background] Mustata S, Groeneveld S, Davidson W, Ford G, Kiland K, Manns B. Effects of exercise training on physical impairment, arterial stiffness and health-related quality of life in patients with chronic kidney disease: a pilot study. Int Urol Nephrol. 2011 Dec;43(4):1133-41. doi: 10.1007/s11255-010-9823-7. Epub 2010 Sep 15. PMID 20842429
- [Background] Goldberg AP, Geltman EM, Gavin JR 3rd, Carney RM, Hagberg JM, Delmez JA, Naumovich A, Oldfield MH, Harter HR. Exercise training reduces coronary risk and effectively rehabilitates hemodialysis patients. Nephron. 1986;42(4):311-6. doi: 10.1159/000183694. PMID 3960242
- [Background] Afshar R, Emany A, Saremi A, Shavandi N, Sanavi S. Effects of intradialytic aerobic training on sleep quality in hemodialysis patients. Iran J Kidney Dis. 2011 Mar;5(2):119-23. PMID 21368391
- [Background] Golebiowski T, Kusztal M, Weyde W, Dziubek W, Wozniewski M, Madziarska K, Krajewska M, Letachowicz K, Strempska B, Klinger M. A program of physical rehabilitation during hemodialysis sessions improves the fitness of dialysis patients. Kidney Blood Press Res. 2012;35(4):290-6. doi: 10.1159/000335411. Epub 2012 Feb 22. PMID 22377500
- [Background] Headley S, Germain M, Mailloux P, Mulhern J, Ashworth B, Burris J, Brewer B, Nindl BC, Coughlin M, Welles R, Jones M. Resistance training improves strength and functional measures in patients with end-stage renal disease. Am J Kidney Dis. 2002 Aug;40(2):355-64. doi: 10.1053/ajkd.2002.34520. PMID 12148109
- [Background] Cheema B, Abas H, Smith B, O'Sullivan A, Chan M, Patwardhan A, Kelly J, Gillin A, Pang G, Lloyd B, Singh MF. Progressive exercise for anabolism in kidney disease (PEAK): a randomized, controlled trial of resistance training during hemodialysis. J Am Soc Nephrol. 2007 May;18(5):1594-601. doi: 10.1681/ASN.2006121329. Epub 2007 Apr 4. PMID 17409306
- [Background] Heiwe S, Jacobson SH. Exercise training for adults with chronic kidney disease. Cochrane Database Syst Rev. 2011 Oct 5;2011(10):CD003236. doi: 10.1002/14651858.CD003236.pub2. PMID 21975737
- [Background] Painter PL, Hector L, Ray K, Lynes L, Dibble S, Paul SM, Tomlanovich SL, Ascher NL. A randomized trial of exercise training after renal transplantation. Transplantation. 2002 Jul 15;74(1):42-8. doi: 10.1097/00007890-200207150-00008. PMID 12134097
- [Background] Boyce ML, Robergs RA, Avasthi PS, Roldan C, Foster A, Montner P, Stark D, Nelson C. Exercise training by individuals with predialysis renal failure: cardiorespiratory endurance, hypertension, and renal function. Am J Kidney Dis. 1997 Aug;30(2):180-92. doi: 10.1016/s0272-6386(97)90051-2. PMID 9261028
- [Background] Padilla J, Krasnoff J, Da Silva M, Hsu CY, Frassetto L, Johansen KL, Painter P. Physical functioning in patients with chronic kidney disease. J Nephrol. 2008 Jul-Aug;21(4):550-9. PMID 18651545
- [Background] Katzmarzyk PT. Physical activity, sedentary behavior, and health: paradigm paralysis or paradigm shift? Diabetes. 2010 Nov;59(11):2717-25. doi: 10.2337/db10-0822. No abstract available. PMID 20980470
- [Background] Rosenberg DE, Norman GJ, Wagner N, Patrick K, Calfas KJ, Sallis JF. Reliability and validity of the Sedentary Behavior Questionnaire (SBQ) for adults. J Phys Act Health. 2010 Nov;7(6):697-705. doi: 10.1123/jpah.7.6.697. PMID 21088299
- [Background] Aaronson NK, Acquadro C, Alonso J, Apolone G, Bucquet D, Bullinger M, Bungay K, Fukuhara S, Gandek B, Keller S, et al. International Quality of Life Assessment (IQOLA) Project. Qual Life Res. 1992 Oct;1(5):349-51. doi: 10.1007/BF00434949. PMID 1299467
- [Background] Studenski S, Perera S, Patel K, Rosano C, Faulkner K, Inzitari M, Brach J, Chandler J, Cawthon P, Connor EB, Nevitt M, Visser M, Kritchevsky S, Badinelli S, Harris T, Newman AB, Cauley J, Ferrucci L, Guralnik J. Gait speed and survival in older adults. JAMA. 2011 Jan 5;305(1):50-8. doi: 10.1001/jama.2010.1923. PMID 21205966
- [Background] Enright PL, McBurnie MA, Bittner V, Tracy RP, McNamara R, Arnold A, Newman AB; Cardiovascular Health Study. The 6-min walk test: a quick measure of functional status in elderly adults. Chest. 2003 Feb;123(2):387-98. doi: 10.1378/chest.123.2.387. PMID 12576356
- [Background] Benzo RP, Sciurba FC. Oxygen consumption, shuttle walking test and the evaluation of lung resection. Respiration. 2010;80(1):19-23. doi: 10.1159/000235543. Epub 2009 Aug 11. PMID 19672050
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Kozey-Keadle S, Libertine A, Staudenmayer J, Freedson P. The Feasibility of Reducing and Measuring Sedentary Time among Overweight, Non-Exercising Office Workers. J Obes. 2012;2012:282303. doi: 10.1155/2012/282303. Epub 2011 Nov 16. PMID 22175004
- [Background] Healy GN, Dunstan DW, Salmon J, Cerin E, Shaw JE, Zimmet PZ, Owen N. Breaks in sedentary time: beneficial associations with metabolic risk. Diabetes Care. 2008 Apr;31(4):661-6. doi: 10.2337/dc07-2046. Epub 2008 Feb 5. PMID 18252901
- [Derived] Lyden K, Boucher R, Wei G, Zhou N, Christensen J, Chertow GM, Greene T, Beddhu S. Targeting Sedentary Behavior in CKD: A Pilot and Feasibility Randomized Controlled Trial. Clin J Am Soc Nephrol. 2021 May 8;16(5):717-726. doi: 10.2215/CJN.12300720. Epub 2021 Apr 22. PMID 33888536
- See also: A 2-Minute Walk May Counter the Harms of Sitting: By Gretchen Reynolds — http://well.blogs.nytimes.com/2015/05/13/a-2-minute-walk-may-counter-the-harms-of-sitting/?_r=0
- See also: . Walking 2 Minutes An Hour Boosts Health, But It's No Panacea. By Patti Neighmond — http://www.npr.org/sections/health-shots/2015/05/01/403523463/two-minutes-of-walking-anhour-boosts-health-but-its-no-panacea
- See also: The Department of Health. The Sedentary Behaviour and Obesity Expert Working Group: Sedentary Behaviour and Obesity: Review of the Current Scientific Evidence — https://www.gov.uk/government/uploads/system/uploads/attachment_data/file/213745/dh_128225.pdf
- See also: Centers for Disease Control and Prevenion. National Center for Health Statistics -NHANES 2003-2004 — http://wwwn.cdc.gov/nchs/nhanes/search/nhanes03_04.aspx
- See also: Utah's Population: Growing fast, Concentrating more, Diversifying rapidly. Utah Legislature Briefing Paper — http://le.utah.gov/lrgc/briefings/PopulationBriefing2014.pdf